CLINICAL TRIAL: NCT02765672
Title: Effectiveness of a Driving Intervention on Safe Community Mobility for Returning Combat Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA Office of Research and Development (U.S. Federal Agency); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201500871; JW 140063 (Other Grant/Funding Number: US Army Med Res and Material Com)
Record Dates: First submitted 2016-05-05; First posted 2016-05-06 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury (TBI); Post Traumatic Stress Disorder (PTSD)
Keywords: Combat Veterans; Automobile Driving; Fitness to Drive
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control Group (Active Comparator): Participants in this group will have the following performed: Institute of Mobility Activity and Participation's clinical battery tests and a simulated driving evaluation, a Brief Driving Behavior Interview, Propensity for Angry Driving Scale, Clinical Driving Assessment, Community Integration Questionnaire, Fitness-to-Drive Screening Measure (FTDS), and a Satisfaction with Life Questionnaire. Driving Safety Education by a traffic safety professional, three x 1 hour sessions to discuss traffic safety rules regarding person, vehicle, environmental factors.
  Interventions: Behavioral: Driving Behavior Interview; Other: Clinical Driving Assessment; Behavioral: Propensity for Angry Driving Scale; Behavioral: Community Integration Questionnaire; Behavioral: Satisfaction with Life; Behavioral: Fitness-to-Drive Screening Measure (FTDS); Procedure: Simulated Driving Evaluation; Procedure: Driving Safety Education
- Experimental Group (Experimental): Participants in this group will have the following performed: Institute of Mobility Activity and Participation's clinical battery tests and a simulated driving tests, a Brief Driving Behavior Interview, Propensity for Angry Driving Scale, Clinical Driving Assessment, Community Integration Questionnaire, Fitness-to-Drive Screening Measure(FTDS), and a Satisfaction with Life Questionnaire. Occupational Therapy Driving Intervention (OT-DI) consisting of three x 1 hour sessions to review explicit driving errors, strategies to mitigate errors and receiving feedback from the evaluator after driving the simulator.
  Interventions: Behavioral: Driving Behavior Interview; Other: Clinical Driving Assessment; Behavioral: Propensity for Angry Driving Scale; Behavioral: Community Integration Questionnaire; Behavioral: Satisfaction with Life; Behavioral: Fitness-to-Drive Screening Measure (FTDS); Procedure: Simulated Driving Evaluation; Procedure: Occupational Therapy Driving Intervention (OT-DI)
- Caregiver Control Group (Active Comparator): Caregiver control group will fill out a Fitness-to-Drive Screening Measure (FTDS) questionnaire at baseline and at the end of the study.
  Interventions: Behavioral: Fitness-to-Drive Screening Measure (FTDS)
- Caregiver Experimental Group (Active Comparator): Caregivers of the experimental group will fill out a Fitness-to-Drive Screening Measure (FTDS) questionnaire at baseline and at the end of the study.
  Interventions: Behavioral: Fitness-to-Drive Screening Measure (FTDS)
- On-road driving Group (Active Comparator): A subset of 30 Combat Veterans will be drawn from the control group (15 no.) and experimental group (15 no.). This group of Combat Veterans will will undergo an on-road driving test at baseline and month 5
  Interventions: Procedure: On-road driving test
- Simulator-drives Evaluation Group (Active Comparator): This group will comprise of 30 Combat Veterans who will be drawn outside of the randomized experimental and and control groups participants. This group will only perform simulator driving triggers evaluation
  Interventions: Procedure: Driving triggers evaluation

INTERVENTIONS:
Behavioral: Driving Behavior Interview — This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test 1)
  Arms: Control Group; Experimental Group
Other: Clinical Driving Assessment — Clinical Driving Assessment includes Optec vision screening, Useful Field of View, Range of Motion, Mini-Mental State Examination (MMSE) and Strength tests. This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test 1)
  Arms: Control Group; Experimental Group
Behavioral: Propensity for Angry Driving Scale — This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test 1)
  Arms: Control Group; Experimental Group
Behavioral: Community Integration Questionnaire — This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test 1)
  Arms: Control Group; Experimental Group
Behavioral: Satisfaction with Life — This will be completed thrice, at baseline, post-test1 and at post-test2 (3 months after post test 1
  Arms: Control Group; Experimental Group
Behavioral: Fitness-to-Drive Screening Measure (FTDS) — Fitness-to-Drive-Screening Measure will be completed twice, at baseline and at end of study
  Arms: Caregiver Control Group; Caregiver Experimental Group; Control Group; Experimental Group
Procedure: Simulated Driving Evaluation — This involves driving a simulator fitted simulated drives engineered to to address Veteran's driving concerns such as reactions to other drivers and road conditions(e.g. debris). The simulator is used at baseline and at post-test1 and 2. The intervention and traffic safety education session 3 also occurs using the driving simulator.
  Arms: Control Group; Experimental Group
Procedure: Driving Safety Education — This involves the following: Session1: general traffic safety discussion; Session 2: Rules of the road and acknowledgement of the road discussion and Session 3: driving the simulator without any feedback from traffic safety professional
  Arms: Control Group
Procedure: Occupational Therapy Driving Intervention (OT-DI) — This has three sessions: 1. Driving evaluator reviews explicit driving errors with Combat Veteran; 2. driving evaluator provide tailored strategies to mitigate errors; Combat Veteran drives simulator with targeted feedback from driving evaluator.
  Arms: Experimental Group
Procedure: On-road driving test — This involves and on-road driving test supervised by Driving Rehabilitation Specialist. To be completed at baseline and at month 5
  Arms: On-road driving Group
Procedure: Driving triggers evaluation — The simulator-drives evaluation group will evaluate the current simulator-triggers prior to baseline testing
  Arms: Simulator-drives Evaluation Group

SUMMARY:
The main objective of this study is to discern if an Occupational Therapy Driving Intervention (OT-DI) improves fitness to drive abilities of Combat Veterans and also investigate if results leads to reduced driving errors on the driving simulator and an on-road test. The driving behavior of 260 Combat Veterans will be studied on a driving simulator at baseline after which they will be randomized into control and intervention groups. The intervention group will receive sessions of Occupational Therapy Driving Intervention by a trained driving rehabilitation specialist. The control group on the other hand will receive driving safety education sessions by a driving safety professional. Both groups will be evaluated for driving performance on the driving simulator to ascertain whether there have been changes in the number of driving errors at two and three months upon enrollment. Caregiver responses on driving behavior of Combat Veteran and public driving records from The Department of Motor Vehicles will be analyzed to for changes in number of driving errors.

DETAILED DESCRIPTION:
This research study is being done to determine if Occupational Therapy Driving intervention (OT-DI) can improve the safe driving performance immediately following intervention and intermediate term (3months).

Baseline testing to post test1 will include Clinical battery of tests and a Simulated Driving test, a Brief Driving Questionnaire, Community Integration Questionnaire, and Satisfaction with Life Questionnaire. Caregivers/family member will rate the participants' driving behaviors using a Fitness-to-Drive Screening Measure (FTDS). After baseline testing the 260 participants (and associated caregivers) will be randomly assigned to balanced intervention and control groups.

The intervention group receives Occupational Therapy Driving Intervention (OT-DI) consisting of three x 1hour sessions will include Sessions1: Driving evaluator reviews explicit driving errors with participants; Session 2: Driving evaluator provides tailored strategies to mitigate errors; Session 3: Participants drive simulator with targeted feedback from driving evaluator.

The control group will receive from a driving safety professional, three x 1 hour general safety sessions (session 1: general traffic safety discussion; Session 2: Rules of the road and acknowledgement of the road discussion; Session 3: drive the simulator without any feedback from a driving safety professional). Immediately after session 3, Post test1 will occur using the same standardized protocol outline for baseline testing.

Post test2: will consist of testing with the same standardized protocol as administered during baseline testing. Caregivers/family members will rate the participants driving behavior using FTDS in addition the investigators will obtain driving data from the Department of Motor Vehicles which include citations, violations, driving mishaps that have occurred for each participant.

To ascertain impact of the OT-DI and driving safety education on real world driving, a subset of 30 participants will be created from the control and intervention groups to perform on-road driving test. The results from this test will be compared with driving performance on the simulated drives.

ELIGIBILITY:
Inclusion Criteria:

* Combat Veterans with polytrauma (mild traumatic brain injury (TBI)/ with accompanying post-traumatic stress disorder (PTSD), traumatic limb amputation/fractures) who drove prior to injury/condition.
* Have a valid driver's license or are eligible for a driver's license.
* Are community dwelling.
* Combat Veterans without formal diagnoses who report driving issues (either formal such as violations, citations or motor vehicle crashes, or informal including risky driving or driving stress and/or anxiety)
* Have potential for following driving safety recommendations Mini-Mental State Examination (MMSE 24/30)
* Are able to participate in a driving evaluation battery.
* Inclusion criterion for caregivers is based on their ability to complete a driving questionnaire pre and post intervention.

Exclusion Criteria:

* Combat Veterans who have severe psychiatric (e.g., psychoses) or physical conditions (e.g., missing both arms and/or legs) that will limit ability to drive;
* Have multiple psychotropic medications that may impact mental or physical (due to side-effects) functioning as per the consulting physician;
* Have severe, un-remediable medical conditions (e.g., severe TBI) as per the consulting physician;
* Pregnant females or those planning pregnancy as determined by self-report.
* Exclusion criterion for caregivers is based on the presence of a cognitive or physical impairment that would hinder their ability to complete the questionnaires or make an active contribution.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Simulator driving errors changes within the experimental and control groups at baseline, months 2 and 5 | Changes in baseline at months 2 and 5
  Simulator driving errors will be quantified at baseline and at month 2 and 5 for the experimental and control groups.

SECONDARY OUTCOMES:
On-road driving errors changes within the experimental and control groups at baseline and month 5 | Changes in baseline at months 5
  Driving errors will be calculated during an on-road test at baseline and at month 5, for the experimental and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sherrilene Classen, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida, Occupational Therapy Department, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No